CLINICAL TRIAL: NCT06200298
Title: Effectiveness of Erector Spinae Plane Block for Percutaneous Arthrodesis of Spinal Fractures: a Randomized Controlled Trial
Brief Title: Effectiveness of Erector Spinae Plane Block for Percutaneous Arthrodesis of Spinal Fractures
Acronym: SPINERECTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020_1299; 2022-A00358-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2023-12-11; First posted 2024-01-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-12

CONDITIONS: SPINAL Fracture; Pain, Postoperative
Keywords: Erector spinae plane block; Spinal trauma; Percutaneous spinal osteosynthesis
MeSH Terms: conditions — Spinal Fractures; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block with naropeine [3,75 mg/mL] (Experimental): Experimental group: Erector spinae plane block with naropeine [3,75 mg/mL]
  Interventions: Procedure: Erector spinae plane block with naropeine [3,75 mg/mL]
- Control group : ESPB with saline 0,9% (Active Comparator)
  Interventions: Procedure: ESPB with saline 0,9%

INTERVENTIONS:
Procedure: Erector spinae plane block with naropeine [3,75 mg/mL] — Erector spinae plane block Procedure:
  * Ultrasound scan with protective sleeve and sterile gel. Research of the thoracic spine process between T8 (for thoracic arthrodesis) and T12 (for lumbar arthrodesis)
  * Once the thorny process is identified, horizontal shift to the transverse process.
  * When the transverse process is spotted, sagittal rotation of the ultrasound probe
  * Skin puncture with an 80 mm hyperechogenic needle in the plane of the ultrasound probe. The needle will be placed in contact with the transverse process
  * Injection, after aspiration, of the solution prepared blindly by the anesthesiologist performing the procedure. For the ESPB group, a long-acting local anaesthetic: ropivacaine 3.75 mg/mL, 30 mL.
  * Repetition of the gesture for the transverse controlateral process
  Arms: Erector spinae plane block with naropeine [3,75 mg/mL]
Procedure: ESPB with saline 0,9% — Procedure for the Erector spinae plane block Procedure by NaCl 0.9%:
  * Ultrasound scan with protective sleeve and sterile gel. Research of the thoracic spine process between T8 (for thoracic arthrodesis) and T12 (for lumbar arthrodesis)
  * Once the thorny process is identified, horizontal shift to the transverse process.
  * When the transverse process is spotted, sagittal rotation of the ultrasound probe
  * Skin puncture with an 80 mm hyperechogenic needle in the plane of the ultrasound probe. The needle will be placed in contact with the transverse process
  * Injection, after aspiration, of the solution prepared blindly by the anesthesiologist performing the procedure. For the control group: saline isotonic serum 30 mL.
  Repetition of the gesture for the transverse controlateral process
  Arms: Control group : ESPB with saline 0,9%

SUMMARY:
Spinal fracture surgery is a common surgery. Post-operative pain has been reduced by the advent of so-called minimally invasive techniques. The immediate post-operative pain, however, remains relatively high, mainly because of muscle pain following the trauma.

The erector spinae plane block (ESPB) is a loco-regional anesthesia technique first described in 2016.

A retrospective cohort study showed an improvement in post-operative analgesia of percutaneous osteosynthesis spinal surgery through a reduction in 24-hour morphine use.

In order to prove and confirm the effectiveness of this technique, we will conduct a double-blind randomized controlled study.

The objective will be to demonstrate the analgesic effectiveness of the technique by reducing morphine consumption in post-operative. The expected reduction in morphine consumption is set at 30%, based on the clinical experience developed in our practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with percutaneous arthrodesis spine surgery for fracture
2. Insured persons
3. Age 18 years
4. Being able to receive informed information
5. Have agreed to participate in writing

Exclusion Criteria:

1. Minor patient
2. Patient refusal
3. Pregnancy
4. Lack of social security coverage
5. Under guardianship or curatorship
6. Inability to express consent
7. History of spinal surgery
8. Unable to use morphine PCA
9. Contraindication to the use of local morphines and/or anesthetics
10. Contraindication to Loco-Regional Anesthesia
11. Long-term opioid patient (Level II and Level III analgesics)
12. Patient with preoperative neuropathic pain (score greater than or equal to 4 on the DN4 questionnaire or taking anti-epileptic or anti-depressant treatments for neuropathic pain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption for the first postoperative 24 hours | during the first 24H after the procedure
  Morphine consumption for the first postoperative 24 hours(mg)

SECONDARY OUTCOMES:
intraoperative morphine consumption | during the procedure
  Post-operative morphic consumption (mg)
Evolution of postoperative morphine consumption 1 hour | Post-operative morphic consumption (mg) at postoperative 1 hour
  Post-operative morphic consumption (mg)
Evolution of postoperative morphine consumption 3 hours | Post-operative morphic consumption (mg) at 3 hours
  Post-operative morphic consumption (mg)
Evolution of postoperative morphine consumption 6 hours | Post-operative morphic consumption (mg) at 6 hours
  Post-operative morphic consumption (mg)
Evolution of postoperative morphine consumption 9 hours | Post-operative morphic consumption (mg) at 9 hours
  Post-operative morphic consumption (mg)
Evolution of postoperative morphine consumption 12 hour | Post-operative morphic consumption (mg) at 12 hours
  Post-operative morphic consumption (mg)
Evolution of postoperative pain | Every 3 hours during the first 24 hours
  Pain evaluation by numerical scale between 0 (none pain) and 10 (worst pain ever)
Duration of stay in postanesthesia care unit (PACU) | when two consecutives Aldrete scores at 10 occure
  Time (minutes) in PACU ; exit criteria = two consecutives Aldrete scores at 10

CONTACTS AND LOCATIONS:
Overall Officials: Cédric CIRENEI, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, Lille, France